CLINICAL TRIAL: NCT00807534
Title: Measurement of Exertional Dyspnea in the Primary Care Setting in Patients With COPD, Phase 2: Sensitivity of the Step Test and Shuttle Walk to Detect Improvement in Dyspnea Following Bronchodilation in Patients With COPD
Brief Title: Sensitivity of New Exercise Tests in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: McGill University (Other); Boehringer Ingelheim (Industry)
Responsible Party: François Maltais, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: BI 244.2513
Record Dates: First submitted 2008-12-10; First posted 2008-12-12 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Exercise; 3-min constant rate stepping test; 3-min constant rate walking test; Bronchodilation; Ipratropium bromide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Ipratropium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ipratropium bromide (Active Comparator): acute bronchodilation: ipratropium bromide
  Interventions: Drug: ipratropium bromide; Behavioral: constant rate step test; Behavioral: constant rate shuttle walk test
- placebo (Placebo Comparator): placebo nebulization
  Interventions: Drug: placebo; Behavioral: constant rate step test; Behavioral: constant rate shuttle walk test

INTERVENTIONS:
Drug: ipratropium bromide — ipratropium bromide nebulization
  Other Names: Atrovent
  Arms: ipratropium bromide
Drug: placebo — placebo nebulization
  Arms: placebo
Behavioral: constant rate step test — nebulization of 500ug
  Other Names: Atrovent
Behavioral: constant rate shuttle walk test — nebulization of 500ug
  Other Names: Atrovent

SUMMARY:
This study was designed to test the following hypothesis:

The 3-min constant rate step test and the 3-min constant rate shuttle walk test will be sensitive to detect improvement in exertional dyspnea following acute bronchodilation in patients with COPD.

DETAILED DESCRIPTION:
BACKGROUND: Cycle and/or treadmill exercise modalities may not adequately reflect the constraints of the physical activities of daily living and may not easily transfer to the primary care setting. Thus, alternatives need to be considered. The use of a continuous shuttle walk test at one or several specified constant walking paces for the assessment of exertional dyspnea has not yet been developed. Since walking is the basic movement for locomotion in everyday life, it seems appropriate to examine the use of a walking test. In addition to walking, one of the most frequent exercise constraints of everyday life lies in the fact of climbing stairs. The step testing methodology has however not specifically focused on the measurement of exertional dyspnea and has not been carried out in patients with COPD. There is a good rationale for the development of a step test for evaluation of exertional dyspnea and exercise tolerance in the primary care setting: (i) simple, inexpensive equipment that requires very little storage space, (ii) ability to externally dictate the work intensity by use of a timing device such as a metronome to regulate the stepping speed, (iii) exercise that is consistent with everyday activity known to be an important dyspnea stimulus (i.e. stair climbing, hill walking), (iv) use of large muscle groups which ensures that ventilation is increased to support the working muscles, with a resultant increase in dyspnea in patients with reduced ventilatory capacity.

GENERAL OBJECTIVE: The general purpose of this investigator-driven initiative is to develop simple exercise tests to assess the effects of pharmacological and rehabilitation interventions on exertional dyspnea in the primary care setting.

METHODS: The study will require five visits at the research centre. The first visit will include pulmonary function testing and an incremental shuttle walking test to characterize the functional capacity of the participants. Patients will also be familiarized to both exercise tests (stepping and walking). The goal of the familiarization will be to reduce the learning effect that typically occurs when an individual completes the same endurance test several times. During the following four visits, patients will complete a total of four exercise tests: two 3-min constant rate step tests and two 3-min constant rate shuttle walks. Each test will be preceded by the nebulization of either a placebo or 500 ug of ipratropium bromide (Atrovent). The placebo or medication will be administered 1 hour prior to the beginning of each test. The study will follow a crossover design, such that each patient will serve as his/her own control. The order of the endurance tests (stepping or walking) will be randomized. Finally, the medication (placebo or ipratropium) will be administered in a randomized, double-blind fashion. The exercise test will be supervised by someone who is unaware of the medication that was administered in order to maintain blinding of the study.

Data analysis: Responsiveness will be evaluated by the change in dyspnea Borg score at completion of the 3-min constant rate stepping test and the 3-min constant rate walking test between the placebo and ipratropium bromide exercises. Paired t tests will be used to evaluate the difference in end-exercise dyspnea between the ipratropium and the placebo conditions for the two forms of exercise. We will also calculate the Standardized Response Mean (SRM), e.g., the mean change in dyspnea Borg score divided by standard deviation (SD) of mean change. A SRM value of 0.5 or more suggests a large change. Bronchodilator-induced changes in E, O2, CO2, and heart rate will be compared between the 3-min constant rate stepping test and the 3-min constant rate walking test. Comparisons will be done using a repeated measure design (ANOVA). Significance level will be set at a p value of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* age > 50 years
* smoking history > 10 packs/year
* post-bronchodilator FEV1 between 30 and 80% predicted and FEV1/FVC < 70% as assessed in previous pulmonary function test (GOLD stage II and III)

Exclusion Criteria:

* respiratory exacerbation within the preceding 2 months
* history of asthma
* significant O2 desaturation (SaO2 < 85%) at rest or during exercise
* presence of another pathology that could influence exercise tolerance

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Dyspnea at the end of the 3-minute walking and stepping exercises | at the end of the 3-minute exercises

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, Principal Investigator — Laval University; Hélène Perrault, Ph.D., Principal Investigator — McGill University
Locations (2):
- Canada (2):
  - Hélène Perrault, Montreal, Quebec
  - François Maltais, Québec, Quebec

REFERENCES:
- [Derived] Sava F, Perrault H, Brouillard C, Darauay C, Hamilton A, Bourbeau J, Maltais F. Detecting improvements in dyspnea in COPD using a three-minute constant rate shuttle walking protocol. COPD. 2012 Aug;9(4):395-400. doi: 10.3109/15412555.2012.674164. Epub 2012 Apr 18. PMID 22509905